CLINICAL TRIAL: NCT01805505
Title: Comparison of Embryo Transfer in Egg Donation Recipients With Transvaginal and Transabdominal Ultrasound
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: slow recruitment rate
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAD-EH-01-2012-01
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Infertility
Keywords: Female infertility; Oocyte donation; Embryo transfer; Transvaginal ultrasonography; Transabdominal ultrasonography
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transvaginal ultrasound-guided embryo transfer (Experimental): Transvaginal ultrasound-guided transfer of two day-3 embryos
  Interventions: Procedure: Transvaginal ultrasound-guided embryo transfer
- Transabdominal ultrasound-guided embryo transfer (Active Comparator): Transabdominal ultrasound-guided transfer of two day-3 embryos
  Interventions: Procedure: Transabdominal ultrasound-guided embryo transfer

INTERVENTIONS:
Procedure: Transvaginal ultrasound-guided embryo transfer — Embryo transfer of two day-3 embryos performed with the Kitazato Long ET catheter (Kitazato Medical Co. Ltd., Tokyo, Japan), guided by transvaginal ultrasound
  Other Names: Kitazato Long ET catheter (Kitazato Medical Co. Ltd., Tokyo, Japan)
  Arms: Transvaginal ultrasound-guided embryo transfer
Procedure: Transabdominal ultrasound-guided embryo transfer — Embryo transfer of two day-3 embryos performed with the Cook Soft-Trans ET catheter (Cook Medical Inc., Bloomington, IN, USA), guided by transabdominal ultrasound
  Other Names: Cook Soft-Trans ET catheter (Cook Medical Inc., Bloomington, IN, USA)
  Arms: Transabdominal ultrasound-guided embryo transfer

SUMMARY:
Transabdominal ultrasound guidance is the golden standard for embryo transfers. Transvaginal ultrasound guidance was proposed recently to provide better visualization and reduce patient discomfort as embryo transfer can be performed with an empty bladder in this case. The purpose of this study is to determine whether there are any differences between transvaginal and transabdominal ultrasound-guided embryo transfer in terms of ease of use, patient satisfaction, and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing oocyte donation treatment with transfer of 2 embryos on day 3

Exclusion Criteria:

* Submucous or >3 cm intramural fibroids
* Turner syndrome
* Black recipients

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 346 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | At performing the pregnancy test 11 days post-embryo transfer
  Proportion of patients with a positive pregnancy test

SECONDARY OUTCOMES:
Clinical pregnancy rate | At first pregnancy ultrasound (3 weeks post-embryo transfer)
  Proportion of patients with at least one gestational sac at first pregnancy ultrasound
Ongoing pregnancy rate | At 10 weeks post-embryo transfer
  Proportion of patients with at least one live intrauterine fetus at 10 weeks post-embryo transfer
Menstruation-like pain | At embryo transfer
  Measured on a three-level scale (none/mild/strong)
Discomfort related to vesical distension | At embryo transfer
  Measured on a three-level scale (none/mild/strong)
Overall discomfort | At embryo transfer
  Measured on a three-level scale (none/mild/strong)
Difficulty using the assigned technique faced by operators | At embryo transfer
  Measured on a three-level scale (easy/moderately difficult/very difficult)
Catheterization time | At embryo transfer
Conversion to the opposite technique | At embryo transfer
  Proportion of cases in which embryo transfer was performed using the technique of the opposite randomization arm (i.e., proportion of patients randomized to have transabdominal ultrasound-guided transfer in whom transvaginal ultrasound-guided was performed, and the other way around)

CONTACTS AND LOCATIONS:
Overall Officials: Erik E Hauzman, MD, PhD, Principal Investigator — IVI Madrid; Juan A Garcia-Velasco, MD, PhD, Study Director — IVI Madrid
Locations (1):
- IVI Madrid, Madrid, Spain